CLINICAL TRIAL: NCT02644291
Title: Phase I Study of Mebendazole Therapy for Recurrent/Progressive Pediatric Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J15211; IRB00072999 (Other: JHMIRB)
Record Dates: First submitted 2015-12-27; First posted 2015-12-31 (Estimated); Last update posted 2022-06-23 (Actual); Status verified 2021-09

CONDITIONS: Medulloblastoma; Astrocytoma, Grade III; Glioblastoma; Anaplastic Astrocytoma; Brain Stem Neoplasms, Malignant; Oligodendroblastoma; Anaplastic Oligodendroglioma; Malignant Glioma
Keywords: medulloblastoma; Diffuse Intrinsic Pontine Glioma (DIPG); high grade glioma; glioblastoma; brain stem malignant glioma
MeSH Terms: conditions — Medulloblastoma; Astrocytoma; Glioblastoma; Brain Stem Neoplasms; Oligodendroglioma; Glioma; Diffuse Intrinsic Pontine Glioma | interventions — Mebendazole; ovex; Piperazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mebendazole (Experimental): oral mebendazole as dose escalation (three groups), or l oral mebendazole at maximum dose for extended cohort. Given in 3 divided doses with meals as chewable 500 mg tablets based on calculated patient surface area.
  Interventions: Drug: Mebendazole

INTERVENTIONS:
Drug: Mebendazole — chewable mebendazole tablets that can also be crushed and mixed with food or drink to be taken daily with meals
  Other Names: Vermox; Ovex; Pripsen

SUMMARY:
This is a safety (Phase 1) trial using mebendazole for recurrent pediatric brain cancers that include medulloblastoma and high grade glioma, that are no longing responding to standard therapies. The drug mebendazole is an oral drug in a chewable 500 mg orange flavored tablet. It is already approved to treat parasitic infections. The purpose of this study is to determine the safety and side effects for increasing doses of mebendazole, followed by the treatment of an additional 12 patients at the best tolerated dose.

DETAILED DESCRIPTION:
The primary objectives of this study are to determine the maximum tolerated dose (MTD) of oral mebendazole in patients with recurrent/progressive pediatric brain tumors and to confirm the tolerance of the MTD of oral mebendazole by assessing tolerance in a dose expansion cohort. Secondary Objectives of the study include to determine the safety, tolerability and toxicity of mebendazole in this patient population, determine the plasma levels of mebendazole in this patient population and Determine progression-free and overall survival of mebendazole in an extended cohort of patients with treatment refractory pediatric brain cancer.

Mebendazole (MBZ) is a drug developed to treat human helminthic disease and is FDA-approved for the treatment of roundworm, common hookworm, American hookworm, pinworm and whipworm. MBZ use is well documented and frequently used in tropical countries at higher doses for the rarer parasitic infections of the brain.

We have shown efficacy in preclinical laboratory models of high grade glioma and medulloblastoma. Mebendazole therapy demonstrated safety in a phase I clinical trial for adults with high grade gliomas such as glioblastoma. This trial completed the maximum approved enrollment of 24 patients treated with mebendazole, with high doses consistent with dosing published for severe parasitic infections.

Laboratory studies indicate that mebendazole enters the brain and brain tumors at concentrations that may be effective for a combination of anti-cancer mechanisms. In animal models of brain cancer evidence suggest that mebendazole can prevent cell proliferation by interfering with tubulin formation, and it may prevent the formation of new abnormal blood vessels that feed tumor growth.

The patients for this experimental trial are those between the age of 1 to 21 with the diagnosis of medulloblastoma, or high grade glioma, where the tumor has resumed growth or continued to grow despite standard medical therapy. High grade glioma are those with a World Health Organization (WHO) grade of III or IV. It includes diagnosis of pediatric glioblastoma, anaplastic astrocytoma, and diffuse intrinsic pontine glioma. Patients who have failed other forms of experimental therapy may also be eligible for this trial.

Mebendazole is provided at no cost in the form of a chewable 500 mg tablets, recommended to be taken three times daily with meals or food. The pill can be chewed after meals, or ground up to be mixed with food or drink. It has a mild orange flavor that is similar in consistency to an antacid tablet.

Although side effects are rare and the vast majority are reversible, they include stomach upset, decreased blood count, and elevated liver enzymes due to inflammation.

The main additional procedure beyond taking this drug, is that patients are requested to consent to up to three additional blood draws to check the blood (serum) levels of the drug to ensure it is being absorbed at sufficient doses.

Patients can continue to receive the drug as long as in the attending physicians opinion the therapy is not causing any severe side effects, and there is no clear indication that the patient will not respond to mebendazole therapy. Patients can withdraw from this trial at any time for any reason, and may be eligible for other experimental therapies afterwards.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a confirmed recurrent/progressive brain malignancy that have failed at least one prior treatment regimen.
2. Age for inclusion in this trial at time of patient enrollment is ≥ 1 year, and up to 21 years (prior to the 22nd birthday) with any of the recurrent medulloblastoma or recurrent high grade glioma may be consented and treated under this protocol. Patients who turn 22 during the course of the trial will continue to be treated.
3. Karnofsky Performance Score (KPS) > 50% for patients ≥10 years of age. Lansky score of ≥ 50 for children < 10 years of age.
4. Life expectancy greater than 10 weeks.
5. Patients must have adequate organ and marrow function as defined below:

   * Leukocytes ≥ 3,000 cells per microliter
   * Absolute Neutrophil Count ≥ 750 cells per microliter
   * Platelets ≥ 75,000 cells per microliter
   * aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal
   * Total Bilirubin < 1.5 x upper limit of normal
   * Creatinine < 1.5 x upper limit of normal OR
   * Creatinine Clearance ≥ 60 mL/min/1.73m2 for patients with creatinine > 1.5 x upper limit of normal
6. The effects of mebendazole on the developing human fetus are unknown. In rats there is evidence of a teratogenic effect, although there is no evidence of adverse effect from women accidently taking mebendazole (at lower doses) during pregnancy. For this reason, women of child-bearing potential should agree to use birth control while taking mebendazole if there is a reasonable risk of pregnancy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
7. Ability for patient (and if applicable parent or legal guardian) understand and the willingness to sign a written informed consent document, or for a parent or legal guardian to give assent for those cases where a very young patient is unable to understand or sign the consent.
8. For the patient or parent/legal guardian to be able to comply with treatment plan, study procedures and follow-up examinations.
9. Failed any previous front line standard of care therapy that is currently used for the patient's initial diagnosis.
10. Ability to swallow pills, or liquid formulation and for patient or parent/legal guardian to keep an accurate medication record.

Exclusion Criteria:

1. Patients who have known allergy to mebendazole.

2 Patients who have previously had a severe side effect, such as agranulocytosis and neutropenia, in conjunction with previous mebendazole or benzimidazole class drug for a parasitic infection.

3 Patients who are taking metronidazole and cannot be safely moved to a different antibiotic greater than 7 days prior to starting mebendazole therapy. Metronidazole and mebendazole in combination have been associated with Stevens-Johnson Syndrome/Toxic Epidermal Necrolysis in a case report.

4 Patients who have previously taken mebendazole as part of any experimental anti-cancer protocol, and have failed this therapy.

5 Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, chronic hepatitis, acute hepatitis, or psychiatric illness/social situation that would limit compliance with study requirements.

6 Pregnant women are excluded because mebendazole is a Class C agent with the potential for teratogenic effects. Because it is not known if mebendazole is excreted in breast milk, breastfeeding should be discontinued if the mother is treated with mebendazole.

7 Patients with human immunodeficiency virus (HIV), hepatitis B surface antigen or hepatitis C positive; or with a history of chronic active hepatitis or cirrhosis.

8 Patients with a history of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risks associated with the study participation or investigational product administration or may interfere with the interpretation of the results.

9 Patients who are not available for follow-up assessments or unable to comply with study requirements.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2016-05; Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Adverse events attributed to mebendazole for patients enrolled in this study | duration of study, approximately two years
  cumulative adverse events from mebendazole therapy in pediatric brain cancer patients

SECONDARY OUTCOMES:
Overall survival for patients enrolled in this study | duration of study , approximately two years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Cohen, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Johns Hopkins University School of Medicine, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Undecided
A peer reviewed publication in a medical journal with the results from the study is planned upon completion of the study,that may/may not have data from individual participants compliant with HIPPA protection.

REFERENCES:
- [Background] Bai RY, Staedtke V, Aprhys CM, Gallia GL, Riggins GJ. Antiparasitic mebendazole shows survival benefit in 2 preclinical models of glioblastoma multiforme. Neuro Oncol. 2011 Sep;13(9):974-82. doi: 10.1093/neuonc/nor077. Epub 2011 Jul 15. PMID 21764822
- [Background] Bai RY, Staedtke V, Rudin CM, Bunz F, Riggins GJ. Effective treatment of diverse medulloblastoma models with mebendazole and its impact on tumor angiogenesis. Neuro Oncol. 2015 Apr;17(4):545-54. doi: 10.1093/neuonc/nou234. Epub 2014 Sep 24. PMID 25253417
- [Background] Bai RY, Staedtke V, Wanjiku T, Rudek MA, Joshi A, Gallia GL, Riggins GJ. Brain Penetration and Efficacy of Different Mebendazole Polymorphs in a Mouse Brain Tumor Model. Clin Cancer Res. 2015 Aug 1;21(15):3462-3470. doi: 10.1158/1078-0432.CCR-14-2681. Epub 2015 Apr 10. PMID 25862759
- [Background] Larsen AR, Bai RY, Chung JH, Borodovsky A, Rudin CM, Riggins GJ, Bunz F. Repurposing the antihelmintic mebendazole as a hedgehog inhibitor. Mol Cancer Ther. 2015 Jan;14(1):3-13. doi: 10.1158/1535-7163.MCT-14-0755-T. Epub 2014 Nov 5. PMID 25376612